CLINICAL TRIAL: NCT04656613
Title: A Phase III, Randomized, Double -Blind, Placebo-controlled Trial to Evaluate Immunogenicity and Safety of the Gam-COVID-Vac Combined Vector Vaccine in Prophylactic Treatment for SARS-СoV-2 Infection in the United Arab Emirates
Brief Title: A Phase III Clinical Trial of the Immunogenicity and Safety of the Gam-COVID-Vac Vaccine Against COVID-19 in the UAE
Acronym: SPUTNIK-UAE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gamaleya Research Institute of Epidemiology and Microbiology, Health Ministry of the Russian Federation (Other)
Collaborators: PDC-CRO (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 06-Gam-COVID-Vac-2020
Record Dates: First submitted 2020-11-30; First posted 2020-12-07 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2020-12

CONDITIONS: Covid19; SARS-CoV Infection
Keywords: vector; covid-19; adenoviral vector vaccine; Sputnik V
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome | interventions — Gam-COVID-Vac vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaccine (Experimental): a study group of 750 subjects receiving the Gam-COVID-Vac combined vector vaccine against the SARS-СoV-2-induced coronavirus infection
  Interventions: Biological: Gam-COVID-Vac
- Placebo (Placebo Comparator): a reference group of 250 subjects receiving placebo
  Interventions: Other: placebo

INTERVENTIONS:
Biological: Gam-COVID-Vac — the Gam-COVID-Vac is combined 2 -component vector vaccine against the SARS-СoV-2-induced coronavirus infection
  Other Names: Sputnik V
  Arms: Vaccine
Other: placebo — Placebo Comparator
  Arms: Placebo

SUMMARY:
This study is randomized, double-blind (blinded for the trial subject and the study physician), placebo-controlled trial in the parallel assignment of the immunogenicity, and safety of the Gam-COVID-Vac combined vector vaccine against the SARS-CoV-2-induced coronavirus infection in adults in the SARS-СoV-2 infection prophylactic treatment.

DETAILED DESCRIPTION:
The subjects will be randomized into two groups in the ratio of 1:3; a reference group of 250 subjects receiving placebo and a study group of 750 subjects receiving the Gam-COVID-Vac combined vector vaccine against the SARS-СoV-2-induced coronavirus infection. The trial subjects will be randomized into five age strata: 18-30, 31-40, 41- 50, 51-60, and 60+ years. Each subject will participate in the trial for 180±14 days after the first dose of the study vaccine/placebo and will have in total six on-site visits to the study physician during the study period and several follow-ups Phone Call/ Teleconsultation during the study as follow:

* One Screening visit, i.e., Screening Visit = Day -7 to Day -1
* Two vaccination visits, i.e.,

  o Visit 1 / Day1
* Tele-consultation / Phone Call to start on Day 2 and a weekly basis until visit 2

  o Visit 2/ Day 21±2 Days
* Tele-consultation / Phone Call to occur on Day 22±2 Days then on a weekly basis until visit 3.
* Four Observational Visits to be scheduled as follow:
* Visit 3/ Day 28 ±2 days
* Weekly Follow Up Tele-consultation / Phone calls until visit 4
* Visit 4/ Day 42 ±4 days
* Weekly Follow Up Tele-consultation / Phone Call until visit 5
* Visit 5/ Day 90 ±7 days
* Weekly Follow Up Tele-consultation / Phone Call until visit 6
* Visit 6/ Day 120 ±14 days
* Weekly Follow Up Tele-consultation / Phone calls until visit 7
* End of Study Visit/ Visit 7/ Day 180 ± 14 days The study vaccine/placebo will be administered intramuscularly during vaccination visits 1 and 2 (day 1 and day 21±2). Subsequent observation visits 3, 4, 5, 6 and end of study visit / EOS /Visit 7 will be made on days 28±2, 42±4, 90±7, 120±14 and D180±14 respectively. During the observation visits, vitals will be assessed in all trial subjects, and changes in the subjects' condition and wellbeing compared to the previous visit will be recorded. Blood samples will be collected per the schedule of assessment from all subjects during the following visits to assess the following immunogenicity parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Agree to sign the study informed consent form (ICF) before performing any study-specific procedure.
2. Adults, i.e., ≥ 18 years old.
3. Negative HIV, hepatitis B, hepatitis C, and syphilis test results
4. Negative IgM and IgG SARS CoV2 antibodies enzyme immunoassay test result.
5. Negative COVID-19 RT-PCR test result at the screening visit.
6. No COVID-19 in medical history.
7. Subjects to confirm they had no contact with COVID-19 persons within at least 14 days before the screening visit.
8. Consent for using effective methods of contraception during the entire trial1
9. A negative urine pregnancy test at the screening visit (for child-bearing age women).
10. Negative alcohol test at the screening visit.
11. No evidence of vaccine-induced reactions or complications after receiving immunobiological products in medical history.
12. No acute infectious and/or respiratory diseases within at least 14 days before the enrollment.

Exclusion criteria:

1. Any vaccination/immunization within 30 days before the enrollment.
2. History of COVID-19.
3. Positive SARS-CoV-2 screening result obtained by PCR (at screening).
4. Test results for IgM and IgG antibodies to SARS-CoV-2 is positive.
5. Administration of steroids (except hormonal contraceptives) and/or immunoglobulins or other blood products therapy not finished 30 days before the enrollment.
6. Pregnancy or breast-feeding.
7. Acute coronary syndrome or stroke suffered less than one year before the enrollment.
8. Tuberculosis, chronic systemic infections in medical history.
9. Drug allergy (anaphylactic shock, Quincke's edema, polymorphic exudative eczema, atopy, serum disease), hypersensitivity or allergic reaction to immunobiological products, known allergic reactions to study vaccine components, acute exacerbation of allergic diseases on the enrollment day.
10. Known allergic reactions to vaccination
11. History of asthma
12. Neoplasms in medical history.
13. Major operations in the past 12 months before study vaccine administration. This will include but not limited to; major organs transplant, bone marrow donation, etc.
14. Splenectomy in the past medical history
15. Neutropenia (absolute neutrophil count <1,000 mm3), agranulocytosis, significant blood loss, severe anemia (hemoglobin <80 g/L), immunodeficiency in the medical history within 6 months before the enrollment.
16. Any family member with immunodeficiency, cancer, or transplantation
17. The active form of a disease caused by the human immunodeficiency virus, syphilis, hepatitis B, or C.
18. Subjects with diabetes, heart disease, chronic kidney disease, or dialysis
19. Subjects with latent tuberculosis infection
20. Anorexia, protein deficiency of any origin.
21. Subjects with any metabolic diseases
22. Tattoos or scars at the injection site (deltoid muscle area), which in the medical opinion of the investigator does not allow assessing the local response to the study vaccine/placebo administration.
23. Alcohol or drug addiction in medical history.
24. Participation in any other interventional clinical trial within the previous 90 days (from the administration of the Vaccine).
25. Any other condition that the study physician considers as a barrier to the trial completion as per the protocol.
26. Healthcare workers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
SARS-CoV-2 glycoprotein-specific antibodies titer | 42±4 , 120±14 and 180±14 days
  The geometric mean titer of the SARS-CoV-2 glycoprotein-specific antibodies in trial subjects on the drug administration day before injecting the first dose of the study vaccine/placebo and 42±4 , 120±14 and 180±14 days after the first dose
Seroconversion rate | 42±4, 120±14 and 180±14 days
  Percentage of trial subjects with fourfold or more increase in the titer of SARS-CoV-2 glycoprotein-specific antibodies in trial subjects on the drug administration day before injecting the first dose of the study vaccine/placebo and 42±4, 120±14 and 180±14 days after the first dose
IFN-gamma antigen-specific release | 28±4 days
  Interferon gamma concentration in response to S protein after re-stimulation with the SARS-CoV-2 glycoprotein in trial subjects on the drug administration day before injecting the first dose of the study vaccine/placebo and 28±4 days after the first dose
CD4+/CD8+ proliferating cells | 28±4 days
  The number of proliferating CD4 and CD8 cells in response to antigen stimulation in trial subjects on the drug administration day before injecting the first dose of the study vaccine/placebo and 28±4 days after the first dose
Virus-neutralizing antibodies titer | 42±4 and 120±14 days
  Geometric mean virus-neutralizing antibodies titer in trial subjects on the drug administration day before injecting the first dose of the study vaccine/placebo and 42±4 and 120±14 days after the first dose

SECONDARY OUTCOMES:
Incidence and severity of adverse events | within 4 & 6 months
  Incidence and severity of adverse events in trial subjects within 4 & 6 months after injecting the first dose of the study vaccine/placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Mostafa, Study Director — PDC-CRO

IPD SHARING:
Plan to Share IPD: No